CLINICAL TRIAL: NCT06307080
Title: Clinical Study of Multimodal Ablation Remodeling Immunosensitized PD-1 in the Treatment of Pancreatic Cancer With Liver Metastasis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiang Long, Chief physician of hepatobiliary and pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023-064
Record Dates: First submitted 2024-02-18; First posted 2024-03-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
Keywords: liver metastases
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-mode thermal ablation combined with intravenous anti-PD-1 and chemotherapy (Experimental): Multimodal ablation therapy +PD-1 antibody combined with intravenous chemotherapy was performed (carreilizumab 200 mg IV D1+ gemcitabine 1000mg/㎡ IV+ albumin binding paclitaxel 125mg/㎡ IV D1.8Q3W; For 6 weeks)
  Interventions: Device: Multi-mode thermal ablation device; Drug: Intravenous anti-PD-1 and chemotherapy
- Intravenous anti-PD-1 and chemotherapy (Active Comparator): Intravenous chemotherapy was performed (carreilizumab 200 mg IV D1+ gemcitabine 1000mg/㎡ IV+ albumin binding paclitaxel 125mg/㎡ IV D1.8Q3W; For 6 weeks)
  Interventions: Drug: Intravenous anti-PD-1 and chemotherapy

INTERVENTIONS:
Device: Multi-mode thermal ablation device — The tumor tissue was rapidly frozen until the ice ball exceeded 5mm of the lesion tissue, kept for 5 minutes, then thawed and warmed. Then, complete ablation was performed according to the radiofrequency temperature control mode of multimodal tumor therapy to ensure that the ablation area included a safe range of 5~10mm around the tumor.
  Arms: Multi-mode thermal ablation combined with intravenous anti-PD-1 and chemotherapy
Drug: Intravenous anti-PD-1 and chemotherapy — intravenous anti-PD-1 and chemotherapy

SUMMARY:
1. Clinical evaluation of multimodal ablation system for pancreatic cancer with hepatic metastatic malignancies.
2. Construction of a combined treatment system of multimodal ablation therapy combined with immunotherapy and chemotherapy.
3. Transformation and clinical application of multimodal ablation system for pancreatic cancer with hepatic metastatic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years old, gender is not limited;
2. Newly diagnosed pancreatic cancer with liver metastasis confirmed by pathology or consistent with clinical diagnosis, and no metastases to organs other than the liver;
3. Imaging evaluable tumors with safe access to puncture;
4. The number of half liver tumors ≤3 and the size of each tumor ≤3 cm;
5. ECOG PS score ≤2 points, expected survival > 3 months.

Exclusion Criteria:

1. Liver function Child-Pugh grade C, severe jaundice, especially obstructive jaundice;
2. The liver is significantly atrophy, the tumor is too large, and the ablation range needs to reach one-third of the liver volume;
3. Expected survival < 3 months;
4. serious heart, lung, liver and kidney dysfunction and coagulation dysfunction;
5. Uncontrolled co-morbidities, including poorly controlled hypertension or diabetes, persistent active infections, or mental illness or social conditions that may affect participants' compliance with the study;
6. refractory ascites, pleural fluid or bad fluid;
7. Pregnancy or breastfeeding;
8. The researcher considers that there are any other factors that are not suitable for inclusion or affect the participant's participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy assessment | Up to 1 year after the treatment
  To evaluate the safety and efficacy of multimodal ablation therapy combined with immunotherapy

SECONDARY OUTCOMES:
Survival benefit | Up to 1 year after the treatment
  Effect on survival benefit of pancreatic cancer patients with liver metastasis

OTHER OUTCOMES:
The application of medical-mechanical combination therapy mode | Up to 1 year after the treatment
  To explore a new combination of drug and device therapy for hepatic metastases of pancreatic cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Long Jiang, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China